CLINICAL TRIAL: NCT03520582
Title: Placement of Novel Endoscopic Enteral Feeding Tube - A Feasibility Study
Brief Title: Placement of Novel Endoscopic Enteral Feeding Tube
Acronym: LEGEND
Status: Terminated | Type: Observational
Why Stopped: stop trial due to proposals for possible optimizations of the device by the investigators.
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 16.22.CLI
Record Dates: First submitted 2016-12-22; First posted 2018-05-11 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers; Enteral Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Volunteers: Cohort of 10 healthy subjects. The tube will be placed and removed by a gastroenterologist experienced in performing endoscopic postpyloric tube placement. Secondly, a second tube will be placed and removed.
  Interventions: Device: Tube placement
- Mechanically ventilated ICU: Cohort of 20 mechanically ventilated intensive care patients requiring a placement of a postpyloric feeding tube on clinical indications.
  Interventions: Device: Tube placement

INTERVENTIONS:
Device: Tube placement — Placement of enteral feeding tubes

SUMMARY:
The aim of this study is to evaluate the technical feasibility of the new tube placement technology in healthy volunteers and, if proven feasible, in critically ill patients requiring placement of a feeding tube.

DETAILED DESCRIPTION:
Enteral feeding is the preferred route of nutrient delivery in hospitalized patients who cannot eat sufficiently. Placement of enteral feeding tubes carries a risk of misplacement especially in patients who are unable to fully collaborate during the tube placement due to neurological impairment and/or the presence of an artificial airway. The misplacement of a feeding tube in the airways has a high risk of severe complications, including pneumonia, mechanical damage of airways and the lung, and death. The verification of correct tube placement can be done using radiography, or interventions aimed at confirming the location of the tube tip by aspiration of gastric contents, and by auscultation during injection of air.

Approximately 20-25 % of patients treated in intensive care units are likely to need placement of a feeding tube, while undergoing mechanical ventilation and having an artificial airway. This high risk patient group would benefit from technologies allowing direct visualization of tube placement. It is also expected that direct visualization of tube placement will allow confirmation of tube placement and therefore eliminate the need of radiography (radiation).

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age >18 years

Patients

* Age >18 years
* mechanically ventilated and requiring a placement of a postpyloric feeding tube on clinical indications
* Informed Consent as documented by signature of relatives

Exclusion Criteria:

Healthy volunteers and patients

* Unrepaired tracheoesophageal fistula
* history of prior esophageal or gastric surgery
* esophageal obstruction, stricture, varices or diverticulum
* esophageal or gastric perforation, gastric or esophageal bleeding
* recent oropharyngeal surgery
* cervical spine injury or anomaly

Additional exclusion criterion for patients only

• know severe coagulopathy (defined as thrombocyte count less than 30x10e9/l or International Normalized Ratio (INR) > 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient in ICU mechanically ventilated and requiring a placement of a postpyloric feeding tube
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Success rate of postpyloric placement, time to reach intragastric and postpyloric position, ease of insertion, handling and image quality. | During Intervention Visit, an average of 24 hours
  using a visual analog scale of 1-10, with 1 indicating the best value

SECONDARY OUTCOMES:
In healthy volunteers, time required to reach gastric and postpyloric placement | During Intervention Visit, an average of 24 hours
  Questionnaire with various positions and the time to reach the position
In healthy volunteers, ease of insertion, handling, and image quality assessed | During Intervention Visit, an average of 24 hours
  Using a visual analog scale of 1-10, with 1 indicating the best value
In healthy volunteers, Usability of specific features - tip steerability, lens rinsing and flushing, air insufflation and fluid extraction | During Intervention Visit, an average of 24 hours
  Using a visual analog scale of 1-10, with 1 indicating the best value.
In patients: Necessity of use of additional sedation/analgesia for the procedure in addition to already established sedation in the context of mechanical ventilation. | During Intervention Visit, an average of 24 hours
  Questionnaire Yes/No and a visual analog scale of 1-10, with 1 indicating the best value
In patients: Ease of insertion, handling, and image quality assessed using a visual analog scale of 1-10, with 1 indicating the best value. | During Intervention Visit, an average of 24 hours
  using a visual analog scale of 1-10, with 1 indicating the best value
In patients: Usability of specific features - tip steerability, lens rinsing and flushing, air insufflation and fluid extraction. | During Intervention Visit, an average of 24 hours
  using a visual analog scale of 1-10, with 1 indicating the best value
In patients: Subjective global assessment of the intensivist on whether or not the technique is suitable for clinical use in patients. | During Intervention Visit, an average of 24 hours
  using a visual analog scale of 1-10, with 1 indicating the best value
In patients: Time required to reach gastric and postpyloric placement | During Intervention Visit, an average of 24 hours
  Questionnaire
In patients: Feasibility of the feeding through Veritract tube. | During Intervention Visit, an average of 24 hours
  using a visual analog scale of 1-10, with 1 indicating the best value
Bleeding and infection related to tube placement | During Intervention Visit, an average of 24 hours
  AE/SAE Questionnaire Yes/No
Erroneous placement in larynx and trachea and associated complications (pneumothorax). | During Intervention Visit, an average of 24 hours
  Outcome mesured with a questionnaire Yes/No
Injuries of the oesophagus, stomach or small intestine related to tube placement. | During Intervention Visit, an average of 24 hours
  Outcome mesured with a questionnaire Yes/No
Reflux of stomach contents during tube placement | During Intervention Visit, an average of 24 hours
  AE/SAE Questionnaire Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Merz, Dr. med., Principal Investigator — Inselspital Bern, Universitätsklinik für Intensivmedizin
Locations (1):
- Universitätsklinik für Intensivmedizin, Bern, Switzerland